CLINICAL TRIAL: NCT05806359
Title: A Randomized, Double-blind, Placebo-controlled, Single Ascending Dose Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Danicamtiv in Healthy Japanese and Caucasian Participants
Brief Title: A Study to Evaluate the Safety, Tolerability, and Drug Levels of Danicamtiv in Healthy Japanese and Caucasian Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CV028-1001
Record Dates: First submitted 2023-03-29; First posted 2023-04-10 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-05

CONDITIONS: Healthy Volunteers
Keywords: Healthy; Danicamtiv; Japanese; Caucasian

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Japanese Cohort - Dose 1 (Experimental)
  Interventions: Drug: Danicamtiv; Drug: Placebo
- Japanese Cohort - Dose 2 (Experimental)
  Interventions: Drug: Danicamtiv; Drug: Placebo
- Japanese Cohort - Dose 3 (Experimental)
  Interventions: Drug: Danicamtiv; Drug: Placebo
- Caucasian Cohort - Dose 3 (Experimental)
  Interventions: Drug: Danicamtiv; Drug: Placebo

INTERVENTIONS:
Drug: Danicamtiv — Specified dose on specified days
  Other Names: BMS-986434; MYK-491
Drug: Placebo — Specified dose on specified days

SUMMARY:
The purpose of this study is to assess the safety, tolerability, and single-dose pharmacokinetics of danicamtiv in healthy Japanese and Caucasian participants.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index between 18 and 30 kilograms/meter squared inclusive, at the screening visit.
* Japanese participants must be of Japanese descent (both biological parents are ethnically Japanese).
* Caucasian participants must be of European or Latin American Caucasian descent.
* A female participant is eligible to participate if she is a woman of nonchildbearing potential as defined in the protocol.
* Males who are sexually active with woman of childbearing potential must agree to follow protocol-defined instructions for method(s) of contraception.

Exclusion Criteria:

* Any acute or chronic medical illness.
* Active infection, including with coronavirus disease-19, diagnosed clinically by the investigator.
* History of any other clinically significant disorder, condition, or disease that, in the opinion of the investigator or sponsor clinical trial physician, would pose a risk to participant safety or interfere with the study evaluation, procedures, or completion.

Note: Other protocol-defined inclusion/exclusion criteria apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2023-03-31 (Actual); Primary Completion 2023-08-14 (Actual); Study Completion 2023-08-14 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events (AEs) | Day 1 up to Day 28
Number of Participants with Vital Sign Abnormalities | Day 1 up to Day 7
Number of Participants with Electrocardiogram (ECG) Abnormalities | Day 1 up to Day 7
Number of Participants with Physical Examination Abnormalities | Day 1 up to Day 7
Number of Participants with Clinical Laboratory Abnormalities | Day 1 up to Day 7

SECONDARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) | Predose and at multiple timepoints (Day 1 up to Day 6) after dosing
Time of Maximum Observed Plasma Concentration (Tmax) | Predose and at multiple timepoints (Day 1 up to Day 6) after dosing
Area Under the Plasma Concentration-time Curve From Time Zero Extrapolated to Infinite Time [AUC(0-inf)] | Predose and at multiple timepoints (Day 1 up to Day 6) after dosing

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Anaheim Clinical Trials, Anaheim, California, United States

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/content/studyconnect/us/en/clinical-trials/NCT05806359.html